CLINICAL TRIAL: NCT06829368
Title: Using Theta-Burst Transcranial Focused Ultrasound Stimulation to Enhance Cognition in Healthy Adults
Brief Title: Transcranial Focused Ultrasound Stimulation to Enhance Cognition in Healthy Participants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Marcus Kaiser, Professor of Neuroinformatics, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: F1558
Record Dates: First submitted 2025-02-05; First posted 2025-02-17 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-02

CONDITIONS: Cognitive Enhancement
Keywords: Transcranial Ultrasound Stimulation; Theta-Burst Stimulation; Cognitive Enhancement; Visual Working Memory; EEG; Mediodorsal Thalamus; Anterior Cingulate Cortex; Anterior Insula; Transcranial Focused Ultrasound Stimulation; Focused Ultrasound Stimulation; Low-Intensity Focused Ultrasound Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: The lateral ventricle is designated as the sham control site, given prior evidence that tFUS targeting this region elicits no detectable effects. This choice facilitates consistent participant expectations across sessions, enabling a reliable baseline comparison. To further reduce bias, participants are blinded to the specific brain region targeted in each session and unaware of whether the stimulation is active or sham. This methodological approach aims to prevent any performance adjustment based on presumed effects of the stimulation, thereby enhancing the validity of the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mediodorsal Thalamus Stimulation (Active Comparator): Theta-burst tFUS targeting the mediodorsal thalamus
  Interventions: Other: Transcranial Focused Ultrasound Stimulation
- Dorsal Anterior Cingulate Cortex Stimulation (Active Comparator): Theta-burst tFUS targeting the dorsal anterior cingulate cortex
  Interventions: Other: Transcranial Focused Ultrasound Stimulation
- Anterior Insula Stimulation (Active Comparator): Theta-burst tFUS targeting the anterior insula
  Interventions: Other: Transcranial Focused Ultrasound Stimulation
- Lateral Ventricle Stimulation (Sham Comparator): Theta-burst tFUS targeting the lateral ventricle.
  Interventions: Other: Transcranial Focused Ultrasound Stimulation

INTERVENTIONS:
Other: Transcranial Focused Ultrasound Stimulation — Using MRI neuronavigation, the investigators will implement theta-burst tFUS in one of the four targets.

SUMMARY:
This study examines the impact of theta-burst transcranial focused ultrasound stimulation (tFUS) on cognitive performance in healthy participants, specifically focusing on both acute and post-stimulation effects on visual working memory (vWM). The investigation will compare TUS effects across targeted deep cortical and subcortical brain regions involved in cognitive processing. Neurophysiological changes following stimulation will be assessed using EEG, providing insight into tFUS-induced modulations in working memory-related brain activity.

DETAILED DESCRIPTION:
This single-blind, crossover trial investigates the effects of theta-burst transcranial focused ultrasound stimulation (tFUS) on visual working memory (vWM) in healthy participants. The study aims to evaluate cognitive enhancement by selectively targeting and comparing three brain structures associated with cognition: (1) the mediodorsal thalamus, (2) the dorsal anterior cingulate cortex, and (3) the anterior insula. Additionally, the lateral ventricle serves as a sham control target.

Each participant will attend four sessions, with each session dedicated to one of the brain structures or the sham site. Sessions consist of three distinct phases: (1) a pre-stimulation phase (task completion prior to tFUS), (2) an on-stimulation phase (task completion concurrent with tFUS), and (3) a post-stimulation phase (task completion following tFUS, with EEG recording). The Object in Place task will be used to assess vWM, requiring participants to recall the colour of abstract objects based on their location or shape.

Primary outcomes focus on both immediate (acute) and delayed (post-stimulation) behavioural changes in task performance, as well as neurophysiological EEG markers indicative of working memory processes. Moreover, the investigators will monitor for immediate and longer-term side effects. Stimulation is administered in a theta-burst pattern for 5 minutes, covering a portion of the task trials during the on-stimulation phase.

This study compares tFUS effects across various deep cortical and subcortical structures, examining acute and post-stimulation cognitive changes and monitoring immediate and longer-term side effects. Findings are expected to offer new insights into the potential of tFUS-based neuromodulation as a tool for cognitive enhancement.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-55years
* Healthy adults with no history of neurological or psychiatric disorders
* Eligible to undergo a T1-weighted MRI scan for tFUS neuronavigational purposes
* Ability to adhere to the tFUS study schedule and complete all assessments
* Right-handed
* Fluent in English
* Abstinence from the use of any recreational drugs in the 48-hour period prior to taking part in the experiment.
* Abstinence from consuming no more than 4 alcoholic units within the 24-hour period before participation.

Exclusion Criteria:

* Any current psychiatric diagnosis
* Neurodevelopmental disorders; history of central nervous system disease, concussion, or other neurological sequelae; presence of tumors, seizures, meningitis, encephalitis, or any abnormal MRI findings of the brain
* Use of any psychotropic medications within five half-lives before the procedure
* Presence of metal implants contraindicated for MRI
* History of head trauma with loss of consciousness
* Calcification in sonicated parts of the brain.
* Visual impairments that cannot be corrected with glasses
* Inability to complete cognitive testing requirements
* Active participation or plans for enrollment in other clinical trials that may impact psychosocial functioning
* History of repeated substance abuse or dependence (excluding nicotine and caffeine); use of medications such as stimulants, modafinil, thyroid medication, or steroids
* No skin disease on or close to the scalp.
* History of seizure or epilepsy; use of medications that lower seizure thresholds
* Claustrophobia or any other condition precluding MRI assessment
* Pregnancy or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Performance Change in Visual Working Memory Task | Measured at three time points (pre-stimulation, on-stimulation, and post-stimulation) during each session. Each participant completes four sessions, occurring once per week over approximately 4 weeks.
  Measuring behavioural change in the modified Object in Place Visual Working Memory task, assessed through accuracy and reaction time.
EEG Changes Post Stimulation | Measured at three time points (pre-stimulation, on-stimulation, and post-stimulation) during each session. Each participant completes four sessions, occurring once per week over approximately 4 weeks.
  Analysis of EEG markers associated with cognitive processes

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Kaiser, Professor of Neuroinformatics, Principal Investigator — University of Nottingham; Mohammad Katshu, Clinical Associate Professor, Principal Investigator — University of Nottingham
Locations (1):
- Neuromodulation Lab, Medical School, Queen's Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided